CLINICAL TRIAL: NCT06637462
Title: DISCRN in Rectal Cancer: DISseCting Response to Neoadjuvant Therapy in Rectal Cancer
Brief Title: A Study of Response to Standard Treatment Before Surgery in People With Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-238
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer; Adenocarcinoma of the Rectum
Keywords: rectal cancer; adenocarcinoma of the rectum; Memorial Sloan Kettering Cancer Center; 24-238
MeSH Terms: conditions — Rectal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Rectal Cancer (Experimental): Participants will be diagnosed with rectal cancer and will be undergoing standard-of-care neoadjuvant therapy.
  Interventions: Diagnostic Test: Endoscopy

INTERVENTIONS:
Diagnostic Test: Endoscopy — Standard of care endoscopy

SUMMARY:
The purpose of the study is to learn more about how the body responds to standard treatment (chemoradiation and chemotherapy). The study will use the results of testing down on participants' blook, tissue, and scans to learn more about how people with rectal cancer respond to chemoradiation and chemotherapy treatment and if it is useful for predicting whether a person's cancer get better, gets worse, or stats the same after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older on day of signing informed consent.
* Have a histologically confirmed diagnosis of invasive adenocarcinoma of the rectum with no known mismatch repair deficiency or Her2 amplification.
* Eligible for and plan to initiate standard-of-care therapy with any of the following regimens:

  * Induction fluoropyrimidine (capecitabine [preferred] or 5-FU) based chemoradiation
  * With plan for consolidative CAPEOX, FOLFOX, or FOLIRINOX
* Woman with childbearing potential who are negative for pregnancy test (urine or blood) and who agree to use an effective contraceptive method. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant. Reliable contraception should be used from the time of screening and must be continued throughout the duration of treatment as per standard of care.

Exclusion Criteria:

* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Patients with prior external beam radiation therapy to the pelvis or brachytherapy seed implantation of the prostate.
* Patients who are pregnant or breastfeeding.
* Men or women not using effective contraception.
* Patients with a contraindication to MR imaging.
* Patients on blood thinners prohibiting endoluminal tumor biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-10-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Up to 3 years
  To define endoscopic (clinical) response to neoadjuvant therapy at the following time points using the MSK regression schema

CONTACTS AND LOCATIONS:
Overall Officials: Paul Romesser, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org